CLINICAL TRIAL: NCT06841276
Title: Evaluation of the Impact of the QoLibri Digital Therapy on Primary Care Patients With Chronic Pain: a Randomized Controlled Clinical Trial.
Brief Title: Impact of QoLibri Medical Device on the Consequences of Chronic Pain: a Randomized Controlled Trial
Acronym: QoLiDoc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Novesia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KM00481
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pain
Keywords: pain, quality of life, functional impact, psychological impact, digital therapy
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QoLibri Digital Therapy (Experimental): Use of the QoLibri Digital Therapy on patient smartphone (on top of Treatment as Usual) for the 6-month experimental phase of the study
  Interventions: Device: QoLibri Digital Therapy
- Wait-list control (No Intervention): Treatment as Usual for the initial 3-month experimental phase (wait list) and then Use of the QoLibri Digital Therapy on patient smartphone for the remaining 3-month experimental phase of the study

INTERVENTIONS:
Device: QoLibri Digital Therapy — A personalized program intended for chronic pain patients. It includes digitalized physical and psychological complementary approaches dedicated to symptoms management and quality of life improvement.
  Arms: QoLibri Digital Therapy

SUMMARY:
A superiority study evaluating the impact of the QoLibri Software as Medical Device on functional and psychological consequences of chronic pain in primary care patients. A prospective, cluster-randomized, wait list, controlled multicentre study with the main objective of evaluating the effectiveness of the QoLibri Digital Therapy on Quality of Life improvement in patients living with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient experiencing at least moderate pain (on the Categorical Pain Scale) for more than 3 months
* Patient with a BPI interference score ≥ 3 in at least 3 out of 7 dimensions
* Patient with a smartphone and an internet connection at the place of use
* Patient affiliated with a social security system or benefiting from such a system

Exclusion Criteria:

* Patient opposing participation in the study
* Patient with severe anxiety and/or depressive disorders (especially a suicidal risk)
* Patient presenting one or more barriers to the initiation of cognitive-behavioral therapy (significant social difficulties, low adherence to current care, insufficient memory or cognitive abilities, lack of time, lack of motivation...),
* Adult patient under legal protection measures (guardianship, legal safeguard, psychiatric care, or deprived of liberty by judicial or administrative decision)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of QoLibri Digital Therapy | month 3
  Pain repercussions measured through the Pain Impact Score (PIS) which combines scores from 3 different domains evaluated by the PROMIS-29 (pain intensity, physical function, and pain interference) and quantifies the extent to which pain interferes with function and daily activities).

SECONDARY OUTCOMES:
Reduction of pain repercussions | day 0, month 3, month 6
  Reduction of pain repercussions measured through the Pain Impact Score (PIS)
Impact on Psychological Health | day 0, month 3, month 6
  Improvement in Mental Quality of Life measured by the MHS score
Impact on Physical Health | day 0, month 3, month 6
  Improvement in Physical Quality of Life measured by the PHS score
Overall Quality of Life | day 0, month 3, month 6
  Improvement in overall Quality of Life measured by the PROMIS-29 domain scores
Global Impression of Change | month 3, month 6
  Evaluation of patient and clinician global impression of change measured by P-GIC and C-GIC
Organizational impact | day 0, month 3, month 6
  Evaluation of care organization measured by an in-house questionnaire
Evaluation of the perceived user experience | month 3, month 6
  Perceived user experience of the patient and the clinician measured by an in-house questionnaire
Evaluation of the perceived severity of pain | day 0, month 3, month 6
  Perceived severity of the pain measured by the Categorical Pain Scale

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Elyn, MD, Principal Investigator
Locations (1):
- Maison de santé Nailloux / Saint-Léon, Nailloux, France

IPD SHARING:
Plan to Share IPD: Undecided